CLINICAL TRIAL: NCT04898387
Title: Efficacy and Safety Assessment of T4030 Eye Drops Versus Ganfort® UD in Ocular Hypertensive or Glaucomatous Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT4030-301
Record Dates: First submitted 2021-05-04; First posted 2021-05-24 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Ocular Hypertension Glaucoma
MeSH Terms: interventions — Ganfort

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The 2 different treatment kits should be identical in external packaging in order to respect the masked evaluation for efficacy and safety.
  The identity of the IMP given to each patient will not be known by the masked investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T4030 Group (Experimental)
  Interventions: Combination Product: Bimatoprost Timolol (T4030)
- Ganfort Group (Active Comparator)
  Interventions: Combination Product: Bimatoprost Timolol (Ganfort)

INTERVENTIONS:
Combination Product: Bimatoprost Timolol (T4030) — Eye drop
  Other Names: Bimatoprost Timolol
  Arms: T4030 Group
Combination Product: Bimatoprost Timolol (Ganfort) — Eye drop
  Other Names: Bimatoprost Timolol
  Arms: Ganfort Group

SUMMARY:
To demonstrate the non-inferiority of T4030 unpreserved eye drops compared to Ganfort® UD in terms of efficacy.

DETAILED DESCRIPTION:
Efficacy Parameters IOP assessment in each eye

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated*
* Patient aged ≥18 years old
* Both eyes with a central corneal thickness assessment ≥500 µm and ≤600 μm a
* Both eyes with diagnosed ocular hypertension or open angle glaucoma

Exclusion Criteria:

* History of narrow angle and/or angle closure glaucoma
* Advanced stage of glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
IOP assessment | Week 12
  The primary efficacy endpoint is the change from Baseline (Day 1) to Week 12 in IOP

SECONDARY OUTCOMES:
Ocular Sign | Week 6 Week 12
  Ocular sign will be assessed through slit lamp examination at each visits

CONTACTS AND LOCATIONS:
Overall Officials: CORENTIN LECAMUS, Study Director — Laboratoires Thea
Locations (1):
- Medical Center Vereya EOOD, Stara Zagora, Bulgaria

IPD SHARING:
Plan to Share IPD: No